CLINICAL TRIAL: NCT02017912
Title: A Phase 2, Randomized, Double Blind, Placebo Controlled Multicenter Study to Evaluate Safety and Efficacy of Transplantation of Autologous Mesenchymal Stem Cells Secreting Neurotrophic Factors (MSC-NTF) in Patients With ALS
Brief Title: Phase 2, Randomized, Double Blind, Placebo Controlled Multicenter Study of Autologous MSC-NTF Cells in Patients With ALS
Acronym: NurOwn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brainstorm-Cell Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BCT-001-US
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Mesenchymal Stromal cells; MSC-NTF; Cell therapy; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurown MSC-NTF cells (Active Comparator): Single autologous MSC-NTF cells treatment by combined intramuscular and intrathecal administration
  Interventions: Biological: Nurown MSC-NTF cells
- Excipient (Placebo Comparator): Combined intramuscular and intrathecal placebo administration
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Nurown MSC-NTF cells — Single autologous MSC-NTF cells treatment by combined intramuscular and intrathecal administration
  Other Names: NurOwn
  Arms: Nurown MSC-NTF cells
Biological: Placebo — Excipient administration by combined intramuscular and intrathecal administration
  Arms: Excipient

SUMMARY:
This is a multi-center, randomized, double blind, placebo controlled study to evaluate the safety and efficacy of autologous (self) transplantation of Neurotrophic factors-secreting Mesenchymal Stromal Cells (MSC-NTF, NurOwn™) in patients with ALS .

MSC-NTF cells are a novel cell-therapeutic approach which is expected to effectively deliver Neurotrophic factors, which are potent survival factors for neurons, directly to the site of damage.

DETAILED DESCRIPTION:
The MSC-NTF cell therapy (NurOwn™) is based on transplantation of autologous bone marrow derived mesenchymal stromal cells (MSC), which are enriched from the patients' own bone marrow, propagated ex vivo and induced to secrete NTFs. The autologous MSC-NTF cells are back-transplanted into the ALS patient into the sites of damage, the spinal cord and the muscles.

NTFs are potent survival factors for embryonic, neonatal, and adult neurons and are considered potential therapeutic candidates for ALS. Delivery of appropriate NTFs to the immediate environment of afflicted neurons in ALS patients is expected to improve their survival and thus slow down disease progression and alleviate symptoms.

Previous open-label clinical trials have shown that MSC-NTF cells treatment was well tolerated and appears to be generally safe. Some initials indications of clinical benefit were also observed in some patients.

This multi-center, randomized, double blind, placebo controlled study will evaluate the safety and efficacy of a single combined intramuscular and intrathecal administration of MSC-NTF cells in early-stage ALS patients. Patients will be followed for approximately three months before transplantation with their autologous MSC-NTF cells or placebo. During this period of time, patient bone-marrow will be harvested and mesenchymal stromal cells will be isolated and expanded. Following treatment patients will be followed for a total of six months at monthly visits.

ELIGIBILITY:
Inclusion Criteria

1. Males and females ages 18 to 75 years old, inclusive.
2. ALS diagnosed as possible, laboratory-supported probable, probable, or definite as defined by revised El Escorial criteria.
3. Disease onset, as defined by first reported occurrence of symptomatic weakness, spasticity, or bulbar symptoms, of more than 12 months and less than or equal to 24 months.
4. Current disease symptoms must include limb weakness.
5. ALSFRS-R ≥30 at the Screening Visit.
6. Upright slow vital capacity (SVC) measure ≥65% of predicted for gender, height, and age at the Screening Visit.
7. Subjects must be taking a stable dose of riluzole for at least 30 days prior to enrolment or not be on riluzole, and not have been on it for at least 30 days prior to enrolment (riluzole-naïve subjects are permitted in the study).
8. Capable of providing informed consent and willing and able to follow study procedures, including willingness to undergo lumbar puncture.
9. Geographic accessibility to the study site and willingness and ability to comply with follow-up.
10. Women of child-bearing potential must agree not to become pregnant for the duration of the study. Women must be willing to consistently use two forms of contraceptive therapy throughout the course of the trial, and undergo a pregnancy test one week before bone marrow aspiration. Men must be willing to consistently use two forms of contraceptive if their partners are of child-bearing age.
11. Citizen or permanent resident of the United States.

Exclusion Criteria:

1. Prior stem cell therapy of any kind.
2. Inability to lie flat for the duration of intrathecal cell transplantation and/or bone marrow biopsy, or inability to tolerate study procedures for any other reason.
3. History of autoimmune disease (excluding thyroid disease) myelodysplastic or myeloproliferative disorder, leukemia or lymphoma, whole body irradiation, hip fracture, or severe scoliosis.
4. Any unstable clinically significant medical condition other than ALS (e.g., within six months of baseline, had myocardial infarction, angina pectoris, and/or congestive heart failure), treatment with anticoagulants that, in the opinion of the investigator, would compromise the safety of patients.
5. Any history of malignancy including any malignancy affecting the central nervous system and melanoma, within the previous 5 years, with the exception of localized skin cancers (with no evidence of metastasis, significant invasion, or re-occurrence within three years of baseline).
6. Serum AST or ALT value >3.0 times the upper normal limit.
7. Serum creatinine value >2.0 times the upper normal limit.
8. Positive test for Hepatitis B, Hepatitis C, HIV.
9. Current use of immunosuppressant medication or use of such medication within 4 weeks of Screening visit (Visit 1).
10. Any history of acquired or inherited immune deficiency syndrome.
11. Exposure to any other experimental agent (off-label use or investigational) or participation in a clinical trial within 30 days prior to Screening Visit (Visit 1).
12. Use of non-invasive ventilation (NIV), diaphragm pacing system or invasive ventilation (tracheostomy).
13. Any history of either substance abuse within the past year, or unstable psychiatric disease according to PI judgment.
14. Placement or usage of feeding tube.
15. Pregnant women or women currently breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merit Cudkowicz, MD, Principal Investigator — Massachusetts General Hospital; Robert H Brown, D.Phil, M.D., Principal Investigator — UMass Medical School; Anthony J. Windebank, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Medical School, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subject population was planned to include up to 48 treated adults, aged 18 to 75 years, with ALS who were randomly assigned (3:1) to the treatment group (36 patients) or placebo group (12 patients). 48 patients were randomized and all 48 patients underwent treatment.
Pre-assignment Details: Visit 1 was the Screening Visit. Visit 2 was the enrollment visit and the pre-transplantation follow-up period (Week 4-6).
  Visit 3 was the second visit of the pre-transplantation follow-up period (Week 8-10), and 1 week before BMA.
  Visit 3, patients were randomized into two arms at a 3:1 ratio. Any patient discontinuing the study prior to transplantation of cells (or placebo) injections was replaced with another subject to meet the target of 48 transplanted patients.
Period: Overall Study
Arm/Group | Nurown MSC-NTF Cells | Excipient
Started | 36 | 12
Completed | 33 | 10
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — miscellaneous | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all participants who were randomized. The FAS was analyzed based upon treatment group subjects were randomized to.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurown MSC-NTF Cells | Excipient | Total
Number analyzed (Participants) | 36 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (11.90) | 53.5 (9.11) | 51.1 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 13
  Male | 25 | 10 | 35
Region of Enrollment [Number; unit: participants]
  United States | 36 | 12 | 48
El Escorial Criteria [Count of Participants; unit: Participants]
  Possible | 3 | 1 | 4
  Laboratory-supported Probable | 5 | 1 | 6
  Probable | 16 | 7 | 23
  Definite | 12 | 3 | 15
ALS Medical History since diagnosis [Mean (Standard Deviation); unit: months] | 9.00 (5.578) | 9.01 (4.637) | 9.00 (5.311)
ALS Medical History since first symptom [Mean (Standard Deviation); unit: months] | 17.62 (3.796) | 16.75 (3.104) | 17.40 (3.624)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least One Treatment Emergent Adverse Events
Description: Safety assessed based on the incidence of treatment-emergent adverse events (TEAEs) (including serious adverse events [SAEs]) including clinically relevant changes in vital signs, clinical laboratory assessments, physical and neurological examinations, and electrocardiogram (ECG) tests, during transplantation of expanded autologous MSC-NTF cells administered on a single occasion via combined intrathecal (IT) administration and intramuscular (IM) injections
Time Frame: Up to 24 weeks following the first intrathecal injection, or End of Study
Population: The safety population includes all randomized participants who receive any study treatment (MSC-NTF or placebo) including those who do not complete the study. The safety population was analyzed based upon the treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Nurown MSC-NTF Cells | Excipient
Number analyzed (Participants) | 36 | 12
Participants | 36 | 12

2. Secondary Outcome: Change in Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R) Slopes From the Pre-transplantation Period to the Post-transplantation Period Between the Treatment and Placebo Groups Through 24 Weeks Post-transplantation.
Description: The ALSFRS-R is a quickly administered (10 minutes) ordinal, validated rating scale (ratings 0-4) used to determine participants' assessment of their capability and independence in 12 functional activities. The total score of ALSFRS-R ranges from 0-48, with higher score being better. The slope of ALSFRS-R for the pre- and post-treatment is obtained from a linear regression model using all available data points in the corresponding period, respectively. The change in slope is obtained from a fixed-effect linear model which is defined as the post-treatment slope minus the pre-treatment slope. The unit of the slope is score on a scale per month. A positive change in slope, means that the patient's decline in the ALSFRS-R score is slower than pre-treatment. A negative change in slope, means that the patient decline in the ALSFRS-R score is faster than pre-treatment.
Time Frame: Up to 24 weeks following the first intrathecal injection
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale per month
Arm/Group | Nurown MSC-NTF Cells | Excipient
Number analyzed (Participants) | 36 | 12
score on a scale per month | -0.556 (0.2784) | -0.356 (0.4821)
Statistical Analysis 1: Comparison: Nurown MSC-NTF Cells vs Excipient; Test type: Superiority; p = 0.7208, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.321 to 0.920], Standard Error of Mean 0.5567

3. Secondary Outcome: Change in SVC Slopes From the Pre-transplantation Period to the Post-transplantation Period Between the Treatment and Placebo Groups Through 24 Weeks Post-transplantation
Description: SVC measures the maximum amount of air exhaled in a single breath, this lung function is influenced by gender, height, and age, in a complex, non-linear, way.
  The SVC reported is a normalized value obtained from a non-linear prediction model that accounts for the influence of participant's gender, height and age.
  SVC was done 3 times at each visit, in order to capture and report the maximal, effort-dependent, lung function that a participant can deliver. The slope of SVC is obtained from a linear regression model using all available data points in the corresponding period, respectively. The change in slope is from a fixed-effect linear model which is defined as the post-treatment slope minus the pre-treatment slope. The unit of the slope is score on a scale per month.
  Positive change in slope, means that the patient's decline in the SVC score is slower than pre-treatment.
  Negative change in slope, means that the patient decline in the SVC score is faster than pre-treatment.
Time Frame: Up to 24 weeks following the first intrathecal injection
Population: The Full Analysis Set (FAS) includes all randomized participants who were randomized. The FAS will be analyzed based upon treatment group subjects were randomized to.
Measure: Least Squares Mean (Standard Error); unit: score on a scale per month.
Arm/Group | Nurown MSC-NTF Cells | Excipient
Number analyzed (Participants) | 36 | 11
score on a scale per month. | -0.73 (0.430) | -0.31 (0.769)
Statistical Analysis 1: Comparison: Nurown MSC-NTF Cells vs Excipient; Test type: Superiority; p = 0.6410, Mixed Models Analysis; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-2.187 to 1.360], Standard Error of Mean 0.881

ADVERSE EVENTS:
Time Frame: From the screening visit through the end of the study period (24 weeks after first treatment)
Description: AE means any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. An AE can be any unfavorable and unintended sign (e.g., an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, without any judgment about causality.
Groups:
- Placebo: Combined intramuscular and intrathecal placebo administration
  Placebo: Excipient administration by combined intramuscular and intrathecal administration
Arm/Group | Nurown MSC-NTF Cells | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/12
Serious Adverse Events (participants affected / at risk) | 8/36 | 1/12
Other Adverse Events (participants affected / at risk) | 36/36 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Nurown MSC-NTF Cells (N=36) | Placebo (N=12)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory fatigue (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 1/11 (1) | 0/2 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Nurown MSC-NTF Cells (N=36) | Placebo (N=12)
Back pain (Musculoskeletal and connective tissue disorders) | 26 (39) | 1 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 17 (27) | 6 (10)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (14) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (13) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (14) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 9 (11) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (10) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 27 (33) | 6 (8)
Muscle contractions involuntary (Nervous system disorders) | 5 (5) | 1 (1)
Paraesthesia (Nervous system disorders) | 5 (6) | 1 (1)
Dysarthria (Nervous system disorders) | 3 (3) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 1 (1)
Balance disorder (Nervous system disorders) | 2 (4) | 0 (0)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Speech disorder (Nervous system disorders) | 2 (2) | 0 (0)
Muscle spasticity (Nervous system disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 26 (78) | 9 (22)
Contusion (Injury, poisoning and procedural complications) | 7 (8) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 7 (8) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (4) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 2 (3) | 2 (2)
Skeletal injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Eye penetration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 19 (20) | 5 (5)
Pyrexia (General disorders) | 12 (12) | 0 (0)
Injection site pain (General disorders) | 10 (10) | 1 (1)
Fatigue (General disorders) | 6 (6) | 1 (1)
Chills (General disorders) | 5 (5) | 0 (0)
Asthenia (General disorders) | 3 (4) | 1 (3)
Feeling hot (General disorders) | 2 (2) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 2 (2) | 1 (1)
Injection site paraesthesia (General disorders) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 1 (2)
Puncture site pain (General disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (12) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (10) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 5 (6) | 2 (3)
Salivary hypersecretion (Gastrointestinal disorders) | 5 (5) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 2 (4) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Erythema induratum (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0)
Grip strength decreased (Investigations) | 2 (2) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 3 (3) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 1/11 (1) | 0/2 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1/11 (2) | 0/2 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-09-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT02017912/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-25): https://cdn.clinicaltrials.gov/large-docs/12/NCT02017912/SAP_001.pdf